CLINICAL TRIAL: NCT05547321
Title: Phase 1 Dose-escalation Trial of OMTX705, an Anti-fibroblast Activation Protein Antibody-drug Conjugate, as Single Agent and in Combination With Anti-PD-1 in Patients With Advanced Solid Tumors
Brief Title: Efficacy and Safety Study of OMTX705, Monotherapy and Anti-PD-1-combined, in Subjects With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oncomatryx Biopharma S.L. (Industry)
Collaborators: Centro de Investigación del Cáncer Universidad de Salamanca (Unknown); CTI Laboratory Services Spain (Unknown); Anapharm Bioanalytics (Unknown); Certara (Industry); Biotrial (Industry); Alcura Health España SA (Unknown); Clinigen, Inc. (Industry); Evidenze (Unknown); TFS Health Science (Unknown); HistoOne (Unknown); Opthimapharm (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OMTX705-001
Record Dates: First submitted 2022-06-02; First posted 2022-09-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — pembrolizumab; Patents as Topic; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Monotherapy (OMTX705) (Experimental): Part 1: OMTX705 is administered as single agent at diffrent escalation doses.
  Interventions: Drug: OMTX705
- Combination (OMTX705 + pembrolizumab) (Experimental): Part 1: OMTX705 at different escalation doses is administered in combination with pembrolizumab at 200 mg.
  Interventions: Drug: OMTX705; Drug: Pembrolizumab
- SARC1 (Experimental): Part 2: OMTX705 is administered as single agent in FAP positive patients at 10 mg/kg
  Interventions: Drug: OMTX705
- PDAC Low (Experimental): Part 2: OMTX705 is administered at 4.0 mg/kg in combination with tislelizumab at 200 mg
  Interventions: Drug: Tislelizumab (BGB-A317); Drug: OMTX705
- PDAC High (Experimental): Part 2: OMTX705 is administered at 7.5 mg/kg in combination with tislelizumab at 200 mg
  Interventions: Drug: OMTX705; Drug: Tislelizumab (BGB-A317)
- SCHED1 (Experimental): Part 2: OMTX705 is administered as single agent at 15 mg/kg
  Interventions: Drug: OMTX705
- BIOPSY (Experimental): Part 2: OMTX705 is administered as single agent at 7.5 mg/kg
  Interventions: Drug: OMTX705

INTERVENTIONS:
Drug: OMTX705 — The investigational product is OMTX705 administered as monotherapy at different escalation doses.
  Arms: Combination (OMTX705 + pembrolizumab); Monotherapy (OMTX705)
Drug: Pembrolizumab — Pembrolizumab at 200 mg administered in combination with different escalation doses of OMTX705.
  Other Names: Keytruda (trademark)
  Arms: Combination (OMTX705 + pembrolizumab)
Drug: OMTX705 — The investigational product is OMTX705 administered as monotherapy at 10 mg/kg
  Arms: SARC1
Drug: OMTX705 — The investigational product is OMTX705 administered as monotherapy at 15 mg/kg
  Arms: SCHED1
Drug: OMTX705 — The investigational product is OMTX705 administered as monotherapy at 7.5 mg/kg
  Arms: BIOPSY; PDAC High
Drug: Tislelizumab (BGB-A317) — Tislelizumab at 200 mg is administered in combination with OMTX705
  Arms: PDAC High; PDAC Low
Drug: OMTX705 — The investigational product is OMTX administered at 4.0 mg/kg
  Arms: PDAC Low

SUMMARY:
Open-label, two parallel arm, multicenter, Phase 1 dose-escalation study to evaluate the safety and tolerability of OMTX705, both as monotherapy or in combination with pembrolizumab (Part 1) or tislelizumab (Part 2) in the treatment of patients with advanced or metastatic cancer in whom there is no available standard therapeutic option.

DETAILED DESCRIPTION:
The study consists of 2 parts:

* Part 1: Phase 1 dose-escalation with two parallel staggered escalation cohorts: one cohort of patients treated with OMTX705 as monotherapy and one cohort of patients receiving escalating doses of OMTX705 in combination with standard pembrolizumab. The combination arm will start once OMTX705 monotherapy safety has been evaluated.
* Part 2: Five cohorts expansions have been projected to confirm the safety of OMTX705 as monotherapy (SCHED1, SARC1 and BIOPSY) and in combination with tislelizumab (PDAC_Low and PDAC_High) will provide additional efficacy and safety information.

For Part 1 (escalation phase) the classical 3+3 design will be followed to establish the maximum tolerated dose (MTD) or the provisional recommended dose for the Part 2 or expansion phase (RP2D). Three to six patients per treatment cohort will be assigned to receive sequentially higher doses of OMTX705 on Days 1 and 8 in cycles of 21 days. The OMTX705 starting dose is 1.0 mg/kg

Dose escalation will be based on a review of all parameters critical to subject safety from C1D1 to the start of C2D1. A safety report will be reviewed by the safty review committee (SRC) to determine if progression to the next planned dose level should occur or if additional subjects or lower dose levels are needed.

Expansion phase (Part 2): Based on the results observed in Part 1, five cohort expansions will provide additional safety and efficacy information and will support the selection of the RP2D and indications to be tested in future efficacy studies.

All patients allocated to receive OMTX705 in combination, will receive the anti-PD-1 tislelizumab. For this particular purpose the following cohorts will be opened:

* Cohort SARC1: OMTX705 in monotherapy at 10 mg/kg in sarcomas expressing FAP with H-score in cancer cells ≥40 or 2+/3+.
* Cohort PDAC_low: OMTX705 at 4.0 mg/kg in combination with tislelizumab in patients with stage IV PDAC.
* Cohort PDAC_high: OMTX705 at 7.5 mg/kg in combination with tislelizumab in patients with stage IV PDAC.
* Cohort SCHED1: Part 1 patient population to receive OMTX705 at 15 mg/kg in monotherapy on Day 1 every 21 days with the possibility to escalate up to 20 mg/kg.
* Cohort BIOPSY: patients with selected indications for which in Part 1 there are hints of antitumor activity who volunteer for paired fresh biopsies. They will receive OMTX705 at 7.5 mg/kg with tislelizumab.

After treatment discontinuation, patients will have the EoT visit 30 (±2) days after the last dose of any component of the treatment for the evaluation of new AEs or recovery from previous ones. EoT visit can be anticipated for patients scheduled to receive the next line of systemic treatment to the day of the start of the new therapy if this happens less than 30 days after the last dose of study treatment.

Subjects who discontinue study treatment for reasons other than progressive disease (PD) will continue to attend PFS Follow-up (FU) Visits every 12 (±1) weeks from the EoT Visit until the occurrence of PD, loss to follow up, consent withdrawal, death, the start of subsequent systemic antineoplastic therapy, or study termination, whichever occurs first.

Only patients enrolled in Part 2 will be followed for survival. To assess survival status, subjects will be contacted (which may be by phone or hospital visit, whichever is preferable) every 3 months from the first dose of OMTX705.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years and older.
2. Part 1 monotherapy and combination: Patients with histologically confirmed advanced (locoregionally recurrent, not amenable to curative therapy) or metastatic solid tumors that have no standard therapeutic option with a proven clinical benefit, or are intolerant to these therapies with any of the following selected tumor histologies: PDAC, gastric cancer (including gastroesophageal junction tumors), head and neck squamous-cell carcinoma (HNSCC), esophageal cancer, NSCLC, high grade serous ovarian cancer, primary peritoneal cancer, mesothelioma, BC, CRC, and FAP positive leiomyosarcoma or other FAP-positive sarcomas (with sponsor's approval). Patients with other tumor histologies may be enrolled with explicit sponsor's approval.

   Part 2:
   * SARC1 cohort: patients with locally advanced or metastatic FAP-positive sarcomas that have no standard therapeutic option with a proven clinical benefit or are intolerant to these therapies. FAP-positive is defined as expression of FAP with an H-score ≥40 or 2+/3+ in a tumor biopsy that can be either archival or fresh. FAP positivity will be considered exclusively on sarcoma cells and not in surrounding fibroblasts or other stromal cells. FAP measurement will be done in a central laboratory provided by the sponsor during the screening period (in countries where this is permitted). Alternatively, eligible patients may have had FAP quantified locally before enrolling the trial as part of the previous care of the patient. In the latter case, FAP will be re-quantified retrospectively in a central lab designated by the sponsor.
   * PDAC_low and_high cohorts: patients with metastatic PDAC who have received at least two and no more than four previous lines of systemic treatment for metastatic disease. If the patient received neoadjuvant/adjuvant therapy and recurred <6 months after the last dose, this line will be counted as the first line for the metastatic disease.
   * SCHED1 cohort: patients with tumors meeting Part 1 definitions.
   * BIOPSY cohort: preferentially patients with metastatic CRC, esophageal cancer, GEJ cancer, gastric or NSCLC that have no standard therapeutic option with a proven clinical benefit or are intolerant to these therapies and volunteer for a fresh pre-treatment biopsy during the screening procedure and on-treatment biopsy. Other tumor histologies can be included after approval from the sponsor´s medical monitor.
3. Patients with tumors with actionable mutations should have progress to all approved and locally available targeted therapies or have them contraindicated.
4. Measurable disease by RECIST 1.1 on computerized tomography (CT), positron emission tomography (FDG-PET) or magnetic resonance (MRI) scan. Imaging tests outside the screening period are valid if performed not more than two weeks before consent signature and otherwise fulfil protocol criteria. In sites where available, FAPI-PET can be used but always with an associated CT.
5. Patients should have documented progression to the last line of therapy or, in the opinion of the investigator, require a change in the therapy. This latter option must be discussed and approved explicitly by the sponsor's medical monitor.
6. ECOG performance status 0-1.
7. Serum albumin ≥3.0 g/dL.
8. Adequate bone marrow, hepatic and renal function:

   1. Total bilirubin ≤1.5 times upper limit of normal (ULN).
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times ULN, (if liver metastases are present, then ≤5 times ULN is allowed).
   3. For Part 1 only: estimated creatinine clearance (CrCL) using the Cockcroft-Gault formula ≥60 mL/minute. Patients with calculated CrCL <60 mL/min can be enrolled if measured CrCL is ≥60 mL/min.
   4. For Part 2 only:, CrCL should be ≥30 mL/min.
   5. Hemoglobin ≥9 g/dL (whole or partial blood transfusions not allowed in the two previous weeks before enrollment).
   6. Absolute neutrophil count (ANC) ≥1.5 x 109/L (growth factors like G-CSF are not allowed in the two previous weeks before enrollment).
   7. Platelet count ≥75 x 109/L (platelet transfusions not allowed in the two previous weeks).
9. Women of childbearing potential (WOCBP) (as defined in Appendix 3) and men with sexual partners who are WOCBP must be willing to adhere to contraceptive requirements as detailed in the protocol (Appendix 3) from at least one month prior to study entry to at least four months after the last dose of study treatment.
10. Suitable venous access for safe drug administration and the study-required drug concentration and PD sampling.
11. For Part 1 only: an archival biopsy for translational research should be available. If the archival biopsy is unavailable or does not have the requirements specified in the sample management plan, it can be replaced with a fresh biopsy. If the archival biopsy is unavailable and the fresh biopsy is not feasible, the medical monitor must approve explicitly the inclusion of the patient. Patients to be enrolled in Part 1 backfilling cohorts should consent for paired screening and on-treatment biopsies.
12. For Part 2 only (Section 6.20.2):

    i.For patients with sarcoma in the cohort SARC1, an archival or fresh biopsy for FAP quantification during the screening period for eligibility is required.

ii.For PDAC_low, PDAC_high and BIOPSY cohorts, the patient must consent for fresh paired biopsies. NOTES: (i) In some exceptional circumstances, the medical monitor can waive the obtention of paired treatment biopsies upon request from the investigator. The rationale for the decision needs to be documented in writing. (ii) A patient receiving treatment can decline the on-treatment biopsy without providing any explanation and continue on study. If it is the investigator who decides to skip the on-treatment biopsy the rationale needs to be discussed with the medical monitor and documented in writing.

iii.For patients enrolled in the SCHED1 cohort, paired fresh biopsies are desirable but voluntary.

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

1. Treatment with systemic anticancer treatments, investigational products, or major surgery within four weeks before the first dose of study drug or five half-lives, whichever is shorter. Subjects should have recovered from previous treatment toxicity to Grade 1, baseline (except alopecia). Patients with endocrinopathies should have the replacement treatment in stable dosing.
2. History of uncontrolled brain metastasis. Subjects with brain metastases are allowed if they are previously treated with surgery, whole-brain radiation, or stereotactic radiosurgery and have new brain imaging confirming that brain metastasis are stable (without evidence of progression by imaging using the identical imaging modality for each assessment, either MRI or CT and considered controlled with <10 mg/day of prednisone-equivalent at the time of receiving the first dose of OMTX705. For asymptomatic subjects, screening brain imaging is not required.
3. Patient has received extended field radiotherapy ≤four weeks before the start of treatment (≤one week for limited field radiation for palliation), and who has not recovered to Grade 1 or better from related side effects of such therapy (except for alopecia).
4. Active infection requiring parenteral or oral antibiotics. Antibiotics given for prophylaxis are allowed. They are also allowed for minor localized infections like cystitis, tonsilitis or localized skin infections.
5. Evidence of a serious uncontrolled medical disorder that, in the opinion of the investigator or medical monitor, makes it unwise for the subject to participate in the study or that might jeopardize compliance with the protocol.
6. Drainage of ascitic or pleural fluid two or more times in the 4 weeks prior to the first dose of study drug or permanent drain in place (e.g, PleurX®) for ascites or pleural effusion symptom management.
7. Psychiatric illness/social circumstances that would limit compliance with study requirements and substantially increase the risk of AEs or compromised ability to provide written informed consent.
8. Clinical evidence of an active second invasive malignancy with the exception of stable prostate cancer on watchful waiting, in situ cervical cancer, breast ductal carcinoma in situ or localized non-melanoma skin cancers.
9. Uncontrolled or significant cardiovascular disease defined by the New York Hearth Association (NYHA) classification III or IV.
10. History of cerebrovascular stroke or myocardial infarction within the previous three months.
11. Grade ≥2 peripheral neuropathy.
12. Baseline QTc (using the Fridericia correction calculation) > 470 msec (unless pacemaker in place, only for patients in Part 2)
13. Combination with pembrolizumab/tislelizumab: history of autoimmune disease requiring systemic immunosuppressive therapy (daily prednisone equivalent doses >10 mg/day).
14. Combination with pembrolizumab/tislelizumab: patients who discontinued prior treatment with any immune checkpoint due to irAEs, irrespective of grade, recovery, or need for continued steroid therapy. Also, subjects without formal contraindication due to previous irAE with any immune checkpoint inhibitor (approved or investigational) are not eligible if the AE has not resolved to Grade 1 or better and/or still requires steroids (>10 mg of prednisone equivalent per day) for ongoing management.
15. Combination with pembrolizumab/tislelizumab: patients with a history of pneumonitis/interstitial lung disease, patients who received live vaccines within 30 days of enrollment, and patients who discontinued prior immune checkpoint inhibitors due to Grade 2 myocarditis are excluded from enrollment into immune checkpoint inhibitor-containing cohorts.
16. Known hepatitis B virus surface antigen seropositive or detectable hepatitis C infection viral load. Note: Subjects who have positive hepatitis B surface antigen antibody can be included but must have an undetectable hepatitis B viral load.
17. Patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must meet the following criteria:

    1. have CD4+ T-cell (CD4+) counts ≥350 cells/μL.
    2. have not had an opportunistic infection within the past 12 months. Patients on prophylactic antimicrobials can be included in the trial.
    3. should be on established antiretroviral therapy for at least four weeks.
    4. have an HIV viral load of less than 400 copies/mL prior to enrollment.
    5. known history of any other relevant congenital or acquired immunodeficiency other than HIV infection.
18. Known or suspected allergy to study treatment or related products, and specifically patients with a prior history of life-threatening reaction to polysorbate 20.
19. Women who are pregnant or breastfeeding or trying to become pregnant.
20. Male patients wishing fathering children, planning for future sperm banking, or expressing concerns about sterility.
21. Patients requiring the concomitant administration of medications that are strong inhibitors or inducers of CYP3A4, 2D6, 1A2, 2C9, 2B6, and 2C19. In case they are taking any of these drugs (Appendix 4), they should be stopped at least 14 days prior to first dose.
22. For Part 1 only: Only in particular circumstances it will be possible to enroll sarcoma patients with negative FAP expression on the surface of the tumor cells (central lab assessment) or without knowing FAP expression levels before C1D1. However, these cases must be discussed and explicitly approved by the sponsor´s medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of OMTX705 | Through study completion, an average of 42 months
  Frequency by grade of treatment-emergent adverse events (TEAEs).

SECONDARY OUTCOMES:
Evaluation of the preliminary signs of antitumor activity of OMTX705 as monotherapy and in combination with pembrolizumab | Through study completion, an average of 42 months
  By assessing the objective response rate (ORR) [complete response (CR) + partial response (PR)] per the Response Evaluation Criteria in Solid Tumors scale version 1.1 (RECIST 1.1)
Evaluation of the OMTX705 Pharmacokinetics | Through study completion, an average of 42 months
  By assessing plasma drug concentrations of OMTX705 as monotherapy and with pembrolizumab/tislelizumab, with Ultra-High-Performance Liquid Chromatography (UPLC-MS/MS) and immunosorbent assay (ELISA) methods
Evaluation of OMTX705 Immunogenicity | Through study completion, an average of 42 months.
  By quantifying the formation of anti-drug antibodies (ADAs) with Meso Scale Discovery (MSD) immunoassay method.

OTHER OUTCOMES:
Evaluation of standard cancer serum biomarkers | Through study completion, an average of 42 months
  By measuring the change in circulating cancer blood biomarkers prior and after using OMTX705 as monotherapy and in combination with pembrolizumab/tislelizumab
Evaluation of OMTX705 biomarkers | Through study completion, an average of 42 months.
  By measuring the changes in circulating OMTX705 biomarkers prior and after using OMTX705 as monotherapy and in combination with pembrolizumab/tislelizumab
Evaluation of OMTX705 payload metabolites | Through study completion, an average of 42 months.
  By quantifying OMTX705 payload TAM470 metabolites prior and after using OMTX705 as monotherapy and in combination with pembrolizumab/tislelizumab.
Evaluation of QTc prolongation | Through study completion, an average of 42 months.
  By performing electrocardiography (ECG) pre and at the end of the OMTX705 infusion as monotherapy and in combination with pembrolizumab/tislelizumab..
Evaluation of cancer-associated fibroblasts (CAFs). | Through study completion, an average of 42 months
  By measuring the changes of CAFs and inmune cells in plasma samples prior and after using OMTX705 as monotherapy and in combination with pembrolizumab.
Evaluation of clinical efficacy of OMTX705 in combination with pembrolizumab/tislelizumab | Through study completion, an average of 42 months
  By assessing the objective response rate (ORR) [complete response (CR) + partial response (PR)] per the Response Evaluation Criteria in Solid Tumors scale version 1.1 (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio García-Ribas, MD, Study Director — Oncomatryx Biopharm, S.L.
Locations (9):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States
- Spain (8):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Universitario de Donostia, San Sebastián, Guipúzcoa
  - Hospital 12 Octubre, Madrid, Madrid
  - Hospital MD Anderson, Madrid, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Onkologikoa, San Sebastián